CLINICAL TRIAL: NCT00662961
Title: Periosteum Versus Bone for the Fixation of Forehead Lift: A Prospective, Randomized, Controlled, Split-Face Trial.
Brief Title: Forehead Lift Fixation
Acronym: Forehead
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Uberlandia (Other)
Responsible Party: Lucas G. Patrocinio, Federal University of Uberlandia
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 2-Patrocinio
Record Dates: First submitted 2008-04-15; First posted 2008-04-21 (Estimated); Last update posted 2008-04-21 (Estimated); Status verified 2008-04

CONDITIONS: Forehead
Keywords: Plastic Surgery

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Periosteum
  Interventions: Procedure: Periosteum
- 2 (Experimental): Bone
  Interventions: Procedure: Bone

INTERVENTIONS:
Procedure: Periosteum — Periosteum fixation
  Arms: 1
Procedure: Bone — Bone tunnel fixation
  Arms: 2

SUMMARY:
To compare periosteum versus bone fixation in forehead lift.

DETAILED DESCRIPTION:
Forehead lift method of fixation is variable and lots of different methods have been described with different rates of success.

The comparison of to different techniques in a RCT has not been reported before.

The objective is to compare periosteum versus bone fixation in forehead lift, in a randomized, blinded, controlled, split-face trial.

ELIGIBILITY:
Inclusion Criteria:

* Eye brow malposition
* Forehead wrinkles

Exclusion Criteria:

* Previous surgery
* Forehead trauma or scar

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2007-01; Primary Completion 2007-07 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Eye brow position | 6 months

SECONDARY OUTCOMES:
Patients' satisfaction | 6 months
Complications | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Lucas G Patrocinio, MD, Principal Investigator — Federal University of Uberlandia, Department of ENT/H&N
Locations (1):
- Federal University of Uberlandia, Department of ENT/H&N, Uberlândia, Minas Gerais, Brazil